CLINICAL TRIAL: NCT05877144
Title: Preservation of Erectile Function With Early Postoperative Application of Low Intensity Shockwave Therapy After Nerve Sparing Radical Prostatectomy
Brief Title: LiSWT for Nerve Sparing Radical Prostatectomy ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2022-0980; JT 22705 (Other: JeffTrial Number)
Record Dates: First submitted 2023-05-05; First posted 2023-05-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Erectile Dysfunction; Localized Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: No Data Available
Masking Description: No Data Available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM I (LiSWT) (Experimental): Patients undergo nerve-sparing radical prostatectomy per standard of care. Patients then receive LiSWT treatment weekly for 6 weeks, then have a 6 week break, followed by 6 more weekly treatments. Patients also undergo DDUS at baseline and during follow up.
  Interventions: Procedure: Nerve-Sparing Prostatectomy; Other: Medical Device Usage and Evaluation; Procedure: Duplex Ultrasound; Other: Survey Administration
- ARM II (sham LiSWT) (Sham Comparator): Patients undergo nerve-sparing radical prostatectomy per standard of care. Patients then receive sham LiSWT treatment weekly for 6 weeks, then have a 6 week break, followed by 6 more weekly treatments. Patients also undergo DDUS at baseline and during follow up.
  Interventions: Procedure: Nerve-Sparing Prostatectomy; Procedure: Sham Intervention; Procedure: Duplex Ultrasound; Other: Survey Administration

INTERVENTIONS:
Procedure: Nerve-Sparing Prostatectomy — Undergo nerve-sparing prostatectomy per standard of care
  Other Names: nerve-sparing radical prostatectomy; nerve-sparing surgery
  Arms: ARM I (LiSWT)
Other: Medical Device Usage and Evaluation — Receive LiSWT
  Arms: ARM I (LiSWT)
Procedure: Duplex Ultrasound — Undergo DDUS
  Other Names: DD; Duplex Doppler; Duplex Doppler Ultrasound
  Arms: ARM I (LiSWT)
Other: Survey Administration — Ancillary studies
  Arms: ARM I (LiSWT)
Procedure: Nerve-Sparing Prostatectomy — Undergo nerve-sparing prostatectomy per standard of care
  Other Names: nerve-sparing radical prostatectomy; nerve-sparing surgery
  Arms: ARM II (sham LiSWT)
Procedure: Sham Intervention — Receive sham LiSWT
  Other Names: Sham Comparator
  Arms: ARM II (sham LiSWT)
Procedure: Duplex Ultrasound — Undergo DDUS
  Other Names: DD; Duplex Doppler; Duplex Doppler Ultrasound
  Arms: ARM II (sham LiSWT)
Other: Survey Administration — Ancillary studies
  Arms: ARM II (sham LiSWT)

SUMMARY:
This phase I clinical trial studies how well low intensity shockwave therapy (LiSWT) improves erectile function in patients who have had nerve-sparing radical prostatectomy (NS-RP), a type of surgery that attempts to save the nerves near the tissues being removed, for prostate cancer. Erectile dysfunction (ED) is a known side effect of the radical prostatectomy procedure. The low intensity shockwave therapy delivers painless electrotherapy pulse to increase blood flow and supply, activation of tissues and wound healing. Using LiSWT after NS-PRP may improve erectile function in men with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether LiSWT following nerve-sparing radical prostatectomy (NS-RP) improves outcomes in men with erectile dysfunction (ED) supported by cGMP phosphodiesterase inhibitor (PDE5i) medication.

SECONDARY OBJECTIVES:

I. To determine whether LiSWT improves duplex doppler ultrasound (DDUS) flow parameters at 6 months following LiSWT treatment.

II. To determine the postoperative durability of any beneficial outcome of LiWST treatment to erectile function.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo nerve-sparing radical prostatectomy per standard of care. Patients then receive LiSWT treatment weekly for 6 weeks, then have a 6 week break, followed by 6 more weekly treatments. Patients also undergo DDUS at baseline and during follow up.

ARM II: Patients undergo nerve-sparing radical prostatectomy per standard of care. Patients then receive sham LiSWT treatment weekly for 6 weeks, then have a 6 week break, followed by 6 more weekly treatments. Patients also undergo DDUS at baseline and during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Men aged 18-80 diagnosed with localized prostate cancer
* Score 12 or higher on the pre-operative International Index of Erectile Function (IIEF) assessment
* Undergo the nerve-sparing radical prostatectomy procedure
* Be taking PDE5i medication for the entirety of the study (normal course of care)
* Be in a sexual relationship with a partner for at least 3 months
* Be willing to attempt sexual activity during the screening period and before each follow-up visit
* Be willing to stop all erectile aids (e.g. prescription and non-prescription erectile medications not part of this study, penile injections, vacuum erection devices, constriction rings) during the screening and study period

Exclusion Criteria:

* • Subject does not speak or understand English

  * Subject has been treated with acoustic wave previously
  * Subject has had prior penile surgery
  * Patients with pacemakers or implantable defibrillators
  * Patients who are using devices which are sensitive to electromagnetic radiation
  * Patients who are found to have metastatic disease and require radiation/hormone therapy before initiation of shockwave/sham treatments
  * Subject has lesions or active infections on the penis or perineum
  * Subject is unwilling to remove piercings from the genital region
  * Subject has a history of substance abuse within 12 months prior, or consuming > 14 alcoholic drinks per week
  * Subject has received an investigational drug within 30 days prior to signing consent
  * Subject has received platelet-rich plasma (PRP) within 3 months of signing consent
  * Subject has received stem cell within 6 months of signing consent
  * Subject has any condition or exhibits behavior that indicates to the principle investigator (PI) that the subject is unlikely to be compliant with study procedures and visits
  * Cognitively/decisionally-impaired individuals

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Patient reported sexual function | At 6 months post low intensity shockwave therapy (LiSWT) initiation
  Will be assessed using the International Index of Erectile Function (IIEF) The IIEF is a15-item questionnaire - each item scored from 0 to 5 - examines five main domains of male sexual function: erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction. Outcomes measured only at 6 months post randomization will be analyzed using analysis of covariance with adjustment for the baseline value.
Patient reported sexual function | At 6 months post low intensity shockwave therapy (LiSWT) initiation
  Will be assessed using the Erection Hardness Scale (EHS). The EHS is a single-item validated Likert scale. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval. Outcomes measured only at 6 months post randomization will be analyzed using analysis of covariance with adjustment for the baseline value.

SECONDARY OUTCOMES:
Change in duplex doppler ultrasound measurement | Baseline to 6 months post LiSWT initiation
  Will be assessed by penile flow parameters. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval. Outcomes measured only at 6 months post randomization will be analyzed using analysis of covariance with adjustment for the baseline value.
Erectile function | At 1 month following LiSWT initiation
  Will be assessed using the IIEF, EHS, Sexual Encounter Profile diary and the Patient Global Impression of Improvement survey scores. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval.
Erectile function | At 3 month following LiSWT initiation
  Will be assessed using the IIEF, EHS, Sexual Encounter Profile diary and the Patient Global Impression of Improvement survey scores. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval.
Erectile function | At 6 month following LiSWT initiation
  Will be assessed using the IIEF, EHS, Sexual Encounter Profile diary and the Patient Global Impression of Improvement survey scores. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval.
Erectile function | At 9 month following LiSWT initiation
  Will be assessed using the IIEF, EHS, Sexual Encounter Profile diary and the Patient Global Impression of Improvement survey scores. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval.
Erectile function | At 12 month following LiSWT initiation
  Will be assessed using the IIEF, EHS, Sexual Encounter Profile diary and the Patient Global Impression of Improvement survey scores. Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, will estimate the mean difference between groups at each time point along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No